CLINICAL TRIAL: NCT06462612
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of Lumateperone in the Acute Treatment of Patients With Manic Episodes or Manic Episodes With Mixed Features Associated With Bipolar I Disorder (Bipolar Mania)
Brief Title: Study of Lumateperone in the Treatment of Patients With Bipolar Mania
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ITI-007-452
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Bipolar Disorder, Manic
MeSH Terms: conditions — Bipolar Disorder | interventions — lumateperone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lumateperone 42 mg (Experimental): Lumateperone 42 mg capsules
  Interventions: Drug: Lumateperone
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lumateperone — Lumateperone 42 mg capsules administered orally, once daily
  Arms: Lumateperone 42 mg
Drug: Placebo — Matching capsules administered orally, once daily
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, study in the acute treatment of patients with a diagnosis of bipolar I disorder with manic episodes or manic episodes with mixed features (bipolar mania), with or without psychotic symptoms, according to criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM 5).

DETAILED DESCRIPTION:
The study will be conducted in 3 phases:

* Screening Period (up to 1 week) during which patient eligibility will be assessed.
* Double-blind Treatment Period (3 weeks) during which all eligible patients will be randomized to receive lumateperone 42 mg or placebo in 1:1 ratio.
* Safety Follow-up Period (1 week) during which all patients will return to the clinic for a safety follow-up visit

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent before the initiation of any study specific procedures;
2. Male or female inpatient, between the ages of 18 and 75 years, inclusive;
3. Meets the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM 5) criteria for bipolar I disorder with a current episode of mania or mania with mixed features with or without psychotic symptoms, as confirmed by a trained and Sponsor-approved rater using the modified Structured Clinical Interview for DSM-5, Clinical Trials Version (SCID-5-CT);
4. YMRS total score ≥ 20 and a score of at least 4 on two of the following YMRS items: irritability, speech, content, and disruptive/aggressive behavior at Screening and Baseline;
5. Hospitalized voluntarily before Screening or admitted to inpatient unit at Visit 1 with a primary diagnosis of mania but not > 14 days before Screening. Hospital admission must be a result of the current manic episode.

Exclusion Criteria:

1. Has a current primary DSM 5 psychiatric diagnosis other than bipolar disorder. These include:

   1. Schizophrenia, schizoaffective disorder, or other psychotic disorders;
   2. Dementia or other cognitive disorders;
   3. Intellectual disability;
   4. Moderate or severe substance use disorder (excluding for nicotine);
2. Experiencing first manic episode;
3. In the opinion of the Investigator, the patient has a significant risk for suicidal behavior during the course of his/her participation in the study or

   1. At Screening, the patient scores "yes" on Items 4 or 5 in the Suicidal Ideation section of the Columbia-Suicide Severity Rating Scale (C-SSRS) within 6 months prior to Screening; or
   2. At Screening, the patient has had 1 or more suicidal attempts within 2 years prior to Screening; or
   3. At Baseline, the patient scores "yes" on Items 4 or 5 in the Suicidal Ideation section of the C-SSRS since the Screening Visit; or
   4. At Screening or Baseline, scores ≥ 4 on Item 10 (suicidal thoughts) on the rater administered Montgomery-Åsberg Depression Rating Scale (MADRS); or
   5. Considered to be an imminent danger to himself/herself or others.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Young Mania Rating Scale (YMRS) | Week 3
  The YMRS is an 11-item, clinician-administered mania rating scale designed to assess the severity of manic symptoms. Four of the YMRS items are rated on a 0 to 8 scale, with the remaining 7 items rated on a 0 to 4 scale. The total score ranges from 0 to 60 with a higher score indicating increased severity of manic symptoms.

SECONDARY OUTCOMES:
Clinical Global Impression Scale-Severity (CGI-S) | Week 3
  The CGI-S is a clinician-rated scale to assess a patient's overall mental health. The scale ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).

CONTACTS AND LOCATIONS:
Locations (31):
- United States (18):
  - Clinical Site, Bentonville, Arkansas
  - Clinical Site, Little Rock, Arkansas
  - Clinical Site, Anaheim, California
  - Clinical Site, Cerritos, California
  - Clinical Site, Orange, California
  - Clinical Site, Torrance, California
  - Clinical Site, Hialeah, Florida
  - Clinical Site, Miami, Florida
  - Clinical Site, Miami Lakes, Florida
  - Clinical Site, Tampa, Florida
  - Clinical Site, West Palm Beach, Florida
  - Clinical Site, Atlanta, Georgia
  - Clinical Site, Stockbridge, Georgia
  - Clinical Site, Chicago, Illinois
  - Clinical Site, Gaithersburg, Maryland
  - Clinical Site, Glen Oaks, New York
  - Clinical Site, Cincinnati, Ohio
  - Clinical Site, Richardson, Texas
- Bulgaria (5):
  - Clinical Site, Burgas
  - Clinical Site, Kazanlak
  - Clinical Site, Plovdiv
  - Clinical Site, Sliven
  - Clinical Site, Sofia
- Romania (3):
  - Clinical Site, Brasov
  - Clinical Site, Bucharest
  - Clinical Site, Iași
- Serbia (5):
  - Clinical Site, Belgrade
  - Clinical Site, Kovin
  - Clinical Site, Kragujevac
  - Clinical Site, Niš
  - Clinical Site, Novi Kneževac

IPD SHARING:
Plan to Share IPD: No